CLINICAL TRIAL: NCT01258504
Title: Influence of Cytochrome P450 3A4 (CYP3A4)-Induction by St. John's Wort (SJW) on the Steady State Pharmacokinetics of Bosentan
Brief Title: Influence of CYP3A4-induction by St. John's Wort on the Steady State Pharmacokinetics of Bosentan
Status: Completed | Type: Observational
Sponsor: Gerd Mikus (Other)
Responsible Party: Sponsor-Investigator, Gerd Mikus, Head of Clinical Research Unit, Heidelberg University
Organization: Heidelberg University (Other)
Other Study IDs: K330; 2010-022328-64 (EudraCT Number)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Drug Interactions
Keywords: Steady-state; Bosentan; St. Johns Wort
MeSH Terms: interventions — Hypericum extract LI 160

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CYP2C9 wild type: CYP2C9 wild type ="extensive metaboliser"
  * Administration of bosentan: 1 x 125 mg p.o. on days 1 and 20, 2 x 62.5 mg p.o. on day 2, 2 x 125 mg p.o. on days 3-19
  * Administration of St. Johns Wort: 3 x 300 mg daily p.o. on days 11-19 and 2 x 300 mg on day 20
  Interventions: Drug: St. Johns Wort
- CYP2C9 mutant: CYP2C9 *2/*2 or 2*/*3 or *3/*3 = "poor metaboliser"
  * Administration of bosentan: 1 x 125 mg p.o. on days 1 and 20, 2 x 62.5 mg p.o. on day 2, 2 x 125 mg p.o. on days 3-19
  * Administration of St. Johns Wort: 3 x 300 mg daily p.o. on days 11-19 and 2 x 300 mg on day 20
  Interventions: Drug: St. Johns Wort

INTERVENTIONS:
Drug: St. Johns Wort — * Administration of bosentan: 1 x 125 mg p.o. on days 1 and 20, 2 x 62.5 mg p.o. on day 2, 2 x 125 mg p.o. on days 3-19.
  * Administration of SJW: 3 x 300 mg daily p.o. on days 11-19 and 2 x 300 mg on day 20
  Other Names: Jarsin

SUMMARY:
The aim of the present study is to assess the impact of the cytochrome P450 2C9 (CYP2C9) genotype (*2 and *3 allele versus wild type; ~3-5% poor metabolisers in Caucasian population) on the pharmacokinetics of bosentan and the impact of CYP3A4-induction by St. John's wort (SJW) on steady state bosentan which is a CYP3A4 inducer itself.

DETAILED DESCRIPTION:
We evaluate the effect of SJW on bosentan pharmacokinetics and its relationship to polymorphisms in the CYP2C9 gene known to reduce CYP2C9 activity. This study will be conducted at bosentan steady-state because concentrations decrease in the first 10 days of treatment due to auto-induction of the metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Good state of health (physically and mentally)
* Able to communicate well with the investigator, to understand and comply with the requirements of the study
* Voluntarily signed informed consent after full explanation of the study to the participant.
* No clinically relevant findings in any of the investigations of the pre-study examination, especially aminotransferase elevations ≥ 3 × upper limit of normal(ULN). Minor deviations of other laboratory values from normal range may be acceptable, if judged by the investigator to be of no clinical relevance.
* Known genotype for CYP2C9 polymorphism.
* Agreement to abstain from alcoholic beverages during the time of the study.
* Females must agree to use a reliable contraception (Pearl Index <1%), e.g. double barrier method.

Exclusion Criteria:

* Any regular drug treatment within the last two months, except for oral contraceptives in female volunteers and L-thyroxine.
* Any intake of a substance known to induce or inhibit drug metabolising enzymes or drug transporters within a period of less than 10 times the respective elimination half-life or 2 weeks, whatever is longer
* Any participation in a clinical trial within the last month before inclusion
* Any physical disorder which could interfere with the participant's safety during the clinical trial or with the study objectives
* Any acute or chronic illness, or clinically relevant findings in the pre-study examination, especially: a) any condition, which could modify absorption, distribution, metabolism, or excretion of the drug regimen under investigation b) Allergies (except for mild forms of hay fever) or history of hypersensitivity reactions
* Regular smoking
* Blood donation within 6 weeks before first study day
* Excessive alcohol drinking (more than approximately 20 g alcohol per day)
* Inability to communicate well with the investigator due to language problems or poor mental development
* Inability or unwillingness to give written informed consent
* Known or planned pregnancy or breast feeding
* Pre-existing moderate or severe liver impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Mikus, Prof. Dr., Principal Investigator — deputy head of department
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Dingemanse J, van Giersbergen PL. Clinical pharmacology of bosentan, a dual endothelin receptor antagonist. Clin Pharmacokinet. 2004;43(15):1089-115. doi: 10.2165/00003088-200443150-00003. PMID 15568889

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosentan: bosentan 125 mg p.o. single dose day 1 bosentan 62.5 mg p.o. b.i.d. day 2-10 bosentan 62.5 mg p.o. b.i.d. day 11-20 SJW 300 mg p.o. t.i.d. day 11-20
Period: Bosentan Single Dose
Arm/Group | Bosentan
Started | 13
Completed | 13
Not Completed | 0
Period: Bosentan Steady-state
Arm/Group | Bosentan
Started | 13
Completed | 13
Not Completed | 0
Period: Bosentan and SJW
Arm/Group | Bosentan
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Bosentan: bosentan 125 mg p.o. day 1 single dose bosentan 62.5 mg p.o. b.i.d. day 2-10 bosentan 62.5 mg p.o. b.i.d. day 11-20 SJW 300 mg p.o. t.i.d. day 11-20
Arm/Group | Bosentan
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Region of Enrollment [Number; unit: participants]
  Germany | 13

OUTCOME MEASURES:

1. Primary Outcome: AUC of Bosentan
Time Frame: 0-infinity; during dosing interval
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/ml
Groups:
- Bosentan After First Dose: bosentan 125 mg p.o. day 1 single dose
- Bosentan at Steady-state: bosentan 62.5 mg p.o. b.i.d. day 2-10
- Bosentan During St John's Wort: bosentan 62.5 mg p.o. b.i.d. day 11-20 SJW 300 mg t.i.d. day 11-20
Arm/Group | Bosentan After First Dose | Bosentan at Steady-state | Bosentan During St John's Wort
Number analyzed (Participants) | 13 | 13 | 13
h*ng/ml | 9540 [7630 to 12000] | 5710 [4530 to 7200] | 5020 [2910 to 8690]

2. Primary Outcome: Cmax of Bosentan
Time Frame: after first dose, at steady-state and during SJW
Measure: Geometric Mean (95% Confidence Interval); unit: ng/ml
Groups:
- Bosentan After First Dose: bosentan125 mg p.o. day 1 single dose
Arm/Group | Bosentan After First Dose | Bosentan at Steady-state | Bosentan During St John's Wort
Number analyzed (Participants) | 13 | 13 | 13
ng/ml | 1620 [1170 to 2240] | 1370 [1050 to 1790] | 1280 [707 to 2300]

ADVERSE EVENTS:
Arm/Group | Bosentan After First Dose | Bosentan at Steady-state | Bosentan During St John's Wort
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 9/13 | 9/13 | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan After First Dose (N=13) | Bosentan at Steady-state (N=13) | Bosentan During St John's Wort (N=13)
feeling of heat (General disorders) | 1 | 0 | 0
headache (General disorders) | 4 | 4 | 1
dyspnea (General disorders) | 1 | 0 | 0
increase of alanine aminotransferase (General disorders) | 1 | 1 | 0
pressure sensation in the head (General disorders) | 1 | 1 | 0
epigastric pressure sensation (General disorders) | 1 | 1 | 0
nasopharyngitis (General disorders) | 1 | 1 | 2
nausea (General disorders) | 1 | 1 | 0
strained muscle (General disorders) | 1 | 1 | 0
nasal congestion (General disorders) | 0 | 0 | 1
ocular itching with secretion of tears (General disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Interindividual changes of the interaction were large suggesting that close monitoring of bosentan effects is advisable because in a sizeable fraction of volunteers the exposure to bosentan was reduced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No